

# Analgesic Effect of Blind Fascia Iliaca Compartment Block Compared to an Ultrasound-guided Femoral Nerve Block in Patients With Hip Fractures

2022-04-26



# **Subject study information**

We would like to ask you to participate in a research project. In this document, you will be informed about the project and what it means to participate.

## What kind of project is this, and why do you want me to participate?

Department responsible for the study is Akutkliniken, Universitetssjukhuset i Linköping, Region Östergötland. Approved by Swedish Ethical Review Authority (Etikprövningsmyndigheten), approval number 2021-05967-01.

## Study title

Analgesic Effect of Blind Fascia Iliaca Compartment Block Compared to an Ultrasound-guided Femoral Nerve Block in Patients With Hip Fractures.

## How will this study be done?

If you have a fracture on the neck of your femur (thigh bone), or high up on the actual femur, and are eligible to receive local anaesthetic near your hip, you will be asked if you would like to participate in this study. It entails us asking you to rate your pain on a scale of 0 to 10, where 10 is the maximum pain, before and 30 minutes after you have received the local anaesthetic.

## Are there any risks?

You will be cared for according to current guidelines, and there will be no difference in your care.

## What happens with the information about me?

The study will collect and register information about you.

Your answers and your results will be handled and processed to prevent unauthorized access. Responsible for your personal details are Erik Müssener, Department director, Akutkliniken, Universitetssjukhuset i Linköping. According to the EU Data Protection Regulation, you have the right to access the information about you that is handled in the study free of charge, and if necessary get any errors corrected. You can also request that the information about you be deleted and that the processing of your personal data be restricted. However, the right to delete and restrict the processing of personal data does not apply when the data is necessary for the research in question. If you want to take part in the information, you must contact Sofia Freland, specialty doctor, Akutkliniken, Universitetssjukhuset i Linköping. The Data Protection Officer can be reached at dataskyddsombud@regionostergotland.se. If you are dissatisfied with how your personal details are processed, you have the right to lodge a complaint with the Privacy Protection Authority (Integritetsskyddsmyndigheten), which is the supervisory authority.

#### How do I get information about the results of the study?

If you wish to receive the results of the study you may contact Sofia Freland, specialty doctor, Akutkliniken, Universitetssjukhuset i Linköping at <a href="mailto:sofia.freland@regionostergotland.se">sofia.freland@regionostergotland.se</a>, or 070-586 86 71.



## **Insurance and compensation**

#### **Participation is voluntary**

Your participation is voluntary and you may choose to cancel your participation at any time. If you choose not to participate or want to cancel your participation, you do not have to state why, nor will it affect your future care or treatment.

If you wish to cancel your participation, please contact the person responsible for the study (see below).

#### Person responsible for the study

Responsible for the study is Sofia Freland, specialty doctor, Akutkliniken, Universitetssjukhuset i Linköping, sofia.freland@regionostergotland.se, 070-586 86 71.



## Consent to participate in the study

I hereby confirm that I have received verbal and/or written information regarding the study "Analgesic Effect of Blind Fascia Iliaca Compartment Block Compared to an Ultrasound-guided Femoral Nerve Block in Patients With Hip Fractures", I have had the opportunity to ask questions. I may keep the written information.

• I consent to participate in the aforementioned study

| Location and date | Participant's signature |
|-------------------|----------------------------|
| | Participant's printed name |